CLINICAL TRIAL: NCT03748875
Title: The Effect of Mindfulness-based Relapse Prevention on Impulsive Control Circuit Among Methamphetamine Dependents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JDu-006
Record Dates: First submitted 2018-10-07; First posted 2018-11-21 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2019-03

CONDITIONS: Methamphetamine-dependence
Keywords: Mindfulness-based relapse prevention; methamphetamine; Prefrontal-striatal circuit; impulsive; mechanism
MeSH Terms: conditions — Impulsive Behavior

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): an 8-session mindfulness-based relapse prevention program
  Interventions: Behavioral: mindfulness-based relapse prevention
- Control group (No Intervention): treatment as usual

INTERVENTIONS:
Behavioral: mindfulness-based relapse prevention — mindfulness-based relapse prevention, 8 weeks
  Arms: Intervention group

SUMMARY:
Amphetamine-type stimulants (ATSs) have become the most important medical issue as well as the social problem. Compared with traditional drugs, ATS are highly neurotoxin and can induce cognitive deficit and psychotic symptoms. Due to lack of efficient medical treatment, psychotherapy and behavioral interventions are the main treatment strategies so far. Mindful-based relapse prevention (MBRP) which combined mindfulness with relapse prevention skills, as a novel intervention, has been widely used in prevent craving and relapse among addictions. While the current research of MBRP mechanism focus on emotion regulation circuit, and there was no study to explore the impulsive circuit, which is the important factor that induce the addiction and relapse. However, there was no report about the influence of MBRP on Prefrontal-striatal circuits. Based on the previous results, the proposed study will focus on evaluating the mechanism of MBRP on prefrontal-striatal circuits, neuropsychological tests and functional MRI will be used to investigate the neurobiological mechanism of MBRP on prefrontal-striatal circuits and related impulsive behaviors.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old, male or female, with 9 years of education or above, can cooperate with the completion of the questionnaire evaluation;
* Comply with DSM-V diagnostic criteria for amphetamine-based addiction;
* The previous use of amphetamines for not less than 1 year (at least once a week);
* Vision and hearing are normal, or in the normal range after correction. No contraindications for magnetic resonance imaging;
* agree to cooperate with the completion of follow-up evaluation;
* The Mindfulness Attention Awareness Scale score is greater than 50 points.

Exclusion Criteria:

* Severe cognitive dysfunction, such as history of head trauma, cerebrovascular disease, epilepsy, etc., drugs used to promote cognitive function in the last 6 months; intellectual impairment IQ<70;
* There have been other abuse or dependence of psychoactive substances in the past 5 years (excluding nicotine); 100 healthy controls have been publicly collected by the public. Exclude serious physical illness and mental damage. through
* SCID clinical interviews exclude family history of mental disorders and psychosis, no history of substance abuse (except nicotine).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
craving change | change from baseline, 4，8，12，27and 52 weeks
  craving will be measured by visual analogue scale(VAS), participants specify their level of craving by indicating a position along a continuous line between two end-points, score ranges from 0 to 10, 0 refers to the lowest level of craving, 10 refers to the highest level of craving
impulsiveness change | baseline，4，8，12，27and 52 weeks
  impulsiveness will be measured by Barratt Impulsiveness Scale, the scale is a 30 item self-report measure, Rarely/Never = 1，Occasionally = 2，Often = 3，Almost Always/Always = 4. Assessment is indicated by the total score added together.
functional connectivity change between prefrontal cortex and striatum | baseline, 8 and 12weeks
  functional connectivity between prefrontal cortex and striatum will be measured by fMRI

SECONDARY OUTCOMES:
cognitive function improvement | baseline，4，8，12，27and 52 weeks
  cognitive function improvement will be measured by Cogstate system
depression level change | baseline，4，8，12，27and 52 weeks
  depression level will be measured by patient health questionnaire-9(PHQ-9). The Patient Health Questionnaire (PHQ) is a multiple-choice self-report inventory, and The PHQ-9 is a tool specific to depression which has 9 items. Assessment is indicated by the total score, which made up by adding together the scores for the scale all seven items.System of scoring is Not at all (0 points),Several days (1 point) More than half the days (2 points) and Nearly every day (3 points).PHQ-9 scores of 5, 10, 15, and 20 represented mild, moderate, moderately severe, and severe depression, respectively.
anxiety level change | baseline，4，8，12，27and 52 weeks
  anxiety level will be measured by Generalized Anxiety Disorder(GAD-7). it has 7 items and measure severity of various signs of GAD according to reported response categories with assigned points. Assessment is indicated by the total score, which made up by adding together the scores for the scale all seven items.System of scoring is Not at all (0 points),Several days (1 point) More than half the days (2 points) and Nearly every day (3 points).
addiction severity change | baseline，4，8，12，27and 52 weeks
  addiction severity will be measured by addiction severity index(ASI). ASI is a semi-structured instrument used in face-to-face interviews conducted by clinicians, researchers or trained techniciansIt measures Medical issues relating to drug use, Employment/Support Status, Levels of Alcohol and Drug Use, Legal Issues Arising from Substance Abuse, Family/Social Factors and Psychiatric/Mental Health Status. Severity ratings are based on the following 10 point scale (0-9).0-1: No real problem, treatment not indicated, 2-3: Slight problem, treatment probably not necessary 4-5: Moderate problem, some treatment indicated 6-7: Considerable problem, treatment necessary 8-9: Extreme problem, treatment absolutely necessary

IPD SHARING:
Plan to Share IPD: Undecided